CLINICAL TRIAL: NCT04733508
Title: Glucagon Like Peptide 1 Receptor (GLP1R) Expression and Beta-cell Mass in Patients With Type 2 Diabetes - the Role of Glucose Homeostasis on Uptake of Beta-cell Tracer Exendin-4
Brief Title: Glucagon Like Peptide 1 Receptor (GLP1R) Expression and Beta-cell Mass in Patients With Type 2 Diabetes
Acronym: GLP1R-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL63933.091.17
Record Dates: First submitted 2020-10-08; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: nuclear imaging; beta cell mass; exendin-4
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 111In-exendin-DTPA (Experimental): Injection of 111In-exendin-DTPA for subsequent localization of the tracer in excised tissue using autoradiography
  Interventions: Drug: 111In-DTPA-exendin-4
- exendin-IRDye800CW (Experimental): Injection of exendin-4-IRDye800CW for subsequent localization of the tracer in excised tissue using fluorescence microscopy
  Interventions: Drug: IRDye800CW-exendin-4

INTERVENTIONS:
Drug: 111In-DTPA-exendin-4 — Injection of 111In-DTPA-exendin-4 and localization of the tracer in excised pancreatic tissue using autoradiography
  Arms: 111In-exendin-DTPA
Drug: IRDye800CW-exendin-4 — Injection of IRDye800CW-exendin-4 and localization of the tracer in excised pancreatic tissue using fluorescence microscopy
  Arms: exendin-IRDye800CW

SUMMARY:
Validation of the exendin-based beta cell imaging technique in patients with type 2 diabetes

DETAILED DESCRIPTION:
Rationale: Reliable imaging biomarkers for non-invasive characterisation of beta-cell mass (BCM) are needed to aid understanding regarding the relationship between beta-cell mass and function during the course of type 2 diabetes (T2D). This study will provide critical information necessary to validate the applicability of exendin-based imaging techniques in patients with T2D. The characterization of beta-cells is currently limited to pancreatic specimens available at autopsy, as in vivo pancreatic biopsy is associated with complications unacceptable in clinical studies. To date, only measurements of circulating C-peptide and insulin levels can be obtained, but these measures do not reflect beta-cell mass, only total beta-cell function. Reliable imaging biomarkers for non-invasive characterisation of beta cell mass are therefore needed. These biomarkers could also be used to validate novel therapeutic strategies aimed to increase or preserve BCM or identify whether patients are eligible for a certain therapeutic strategy (e.g. when certain amount of beta-cells is required). One can also think of identifying early responders to therapies, to avoid unnecessary drug use and the accompanying costs.

The objective of this study is to determine the specificity of Exendin-4 during the course of T2D and to examine the role of glycemic control on the correlation between pancreatic Exendin-4 uptake, BCM and GLP-1R expression in patients with T2D undergoing (partial) pancreatectomy. This will allow examination of the role of glycemic control on exendin uptake in humans, but also implementation of clinical guidelines for the interpretation of clinical exendin-based scans in patients with T2D to avoid false interpretation of the scans.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for partial or complete pancreatectomy at Radboudumc

Exclusion Criteria:

* Previous treatment with synthetic exendin or dipeptidyl-peptidase IV inhibitors within the past 3 months
* Breast feeding
* Pregnancy or the wist to become pregnant within 6 months
* Creatinine clearance below 40ml/min
* Liver disease defined as aspartate aminotransferase of alanine aminotransferase level of more than three times the upper limit of normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic exendin uptake 111In-DTPA exendin-4 | 111In-DTPA-exendin-4 injection will be performed a day before planned surgery, and uptake will be determined using ex vivo SPECTof the resected tissue one day after surgery
  The pancreatic uptake of 111In-DTPA-exendin-4 will be quantified using ex vivo SPECT
Pancreatic exendin uptake 111In-DTPA exendin-4 | 111In-DTPA-exendin-4 injection will be performed a day before planned surgery, and uptake will be determined with tissue autoradiography immediately after resection
  The pancreatic uptake of 111In-DTPA-exendin-4 will be quantified using tissue autoradiography
Beta cell function | The glucose tolerance test will be performed within a week before planned surgery
  The beta cell function will be determined with a glucose tolerance test
Blood glucose levels | Blood glucose levels will be continuously monitored a week prior to surgery
  Glycemic control will be determined by monitoring blood glucose levels
HbA1C levels | HbA1C levels will be determined within a week before planned surgery
  HbA1C levels will be determined as a measure of glycemic control
Pancreatic exendin uptake IRDye800CW-exendin-4 | IRDye800CW-exendin-4 injection will be performed a day before planned surgery, and uptake will be determined using microscopy in the excised tissue
  Uptake of IRDye800CW-exendin4 will be visualized with microscopy
Gene expression | Gene expression will be determined in the excised pancreatic tissue immediately after resection
  Gene expression levels will be determined with quantitative polymerase chain reaction (qPCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jansen TJP, Tokgoz S, Buitinga M, van Lith SAM, Joosten L, Frielink C, Smeets EMM, Stommel MWJ, van der Kolk MB, de Galan BE, Brom M, Boss M, Gotthardt M. Validation of radiolabelled exendin for beta cell imaging by ex vivo autoradiography and immunohistochemistry of human pancreas. EJNMMI Res. 2024 Oct 15;14(1):96. doi: 10.1186/s13550-024-01159-6. PMID 39405026